CLINICAL TRIAL: NCT06712576
Title: Evaluation of Planned Conservative Surgical Management of Placenta Accreta Spectrum in Women's Health Center, Assiut University Hospital
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Gamal Ahmed Saleh, resident doctor Obsetitric and Gynacology, Assiut University
Other Study IDs: placenta accreta spectrum
Record Dates: First submitted 2024-11-27; First posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Placenta Accreta
Keywords: planned conservative surgical managemen
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with placenta accrete spectrum: patients with placenta accrete spectrum secondary to previous cesarean section will be recruited from the outpatient clinic and reception unit, Assiut, Egypt.

SUMMARY:
In recent years, with the application of an abdominal artery balloon and the improvement of surgical techniques, efforts are made to preserve the uterus for patients PAS. the aim of the study To evaluate conservative surgical management of placenta accreta spectrum in Assiut University hospital regarding maternal and fetal outcomes.

DETAILED DESCRIPTION:
Placenta accreta spectrum disorder (PAS) is a serious obstetric disorder that is characterized by low lying and deep penetration of the villi which are abnormally attached to the myometrium of the uterus. This obstructs its complete separation during the third stage of labor which induces continued bleeding and have potentially life- threatening for the mother. Most commonly, it is a consequence of a partial or complete absence of the compact and spongy layer known as the decidua basalis, and mis-development of the fibrinoid Nitabuch's layer which lies between the boundary zone of the thick endometrium and the cytotrophoblastic shell in the placenta.

Traditionally, caesarean hysterectomy at the time of delivery has been the preferred management strategy for placenta previa accreta. Not only does this approach preclude future fertility, but it is also a procedure synonymous with significant perioperative risks. For women who wish to conserve their reproductive function, other treatment options have been described.

Different methods have been employed to manage the PA, ranging from uterine conservation, which involves leaving the placenta in situ, to conventional hysterectomy. Classical cesarean sections (C- sections) prevent the excessive bleeding by leaving the adherent placenta in situ and by adopting strategic planning with a comprehensive analysis that aids the reduction in maternal morbidity and mortality rates.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women with history of previous caesarean section.
2. Age above 18 years.
3. Gestational age above 28 weeks.
4. U/S signs suggestive of placenta previa accreta.
5. Confirmed diagnosis of Placenta previa accreta spectrum disorder by 3 D U/S, Doppler or MRI if needed.

Exclusion Criteria:

1. Gestational age less 28 weeks.
2. Age less than 18 years.
3. Patients with known bleeding disorders.
4. Multiple pregnancy.
5. Other pathology (fibroid, ………………..).
6. Patients with placental separation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Study Population: patients with placenta accrete spectrum secondary to previous cesarean section and Gestational age above 28 weeks
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
amount of blood loss | baseline
  amount of blood loss during operation according to number of towels and amount of blood in suction pump

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Cali G, Forlani F, Giambanco L, Amico ML, Vallone M, Puccio G, Alio L. Prophylactic use of intravascular balloon catheters in women with placenta accreta, increta and percreta. Eur J Obstet Gynecol Reprod Biol. 2014 Aug;179:36-41. doi: 10.1016/j.ejogrb.2014.05.007. Epub 2014 May 21. PMID 24965977